CLINICAL TRIAL: NCT01638975
Title: Testing the Feasibility of Response Inhibition Enhancement Training for Individuals With Trichotillomania
Brief Title: Response Inhibition Training for Individuals With Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Trichotillomania Learning Center (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLC 2010 Lee
Record Dates: First submitted 2012-06-16; First posted 2012-07-12 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Trichotillomania
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized response inhibition training (Experimental): Participants in this condition receive 8 computerized training sessions over a 4 week period.
  Interventions: Behavioral: Response Inhibition Training Program
- Waitlist Control (No Intervention): Participants assigned to this condition wait without an intervention until the second assessment (4 weeks after the baseline assessment).

INTERVENTIONS:
Behavioral: Response Inhibition Training Program — This is a computerized cognitive retraining program consisting of 8 sessions delivered over a 4-week period.
  Arms: Computerized response inhibition training

SUMMARY:
This study tests a computerized cognitive training program designed for young individuals with compulsive hair pulling (also known as trichotillomania;TTM). Research suggests that individuals with TTM are characterized by poor cognitive abilities to suppress irrelevant response. This ability is called response inhibition. The current study tests a cognitive training program designed to improve individuals' cognitive abilities of response inhibition through a 8-session computerized training program. The investigators hypothesize that those who complete the response inhibition training program will show a greater reduction in hair pulling symptoms, compared to those assigned to a waitlist group.

DETAILED DESCRIPTION:
Despite ongoing research into causes and treatments for trichotillomania, it remains poorly understood, underdiagnosed and inadequately treated. Further, treatment of TTM in children has received little attention, and only recently have the investigators begun to see research in pediatric trich. One possible way of progressing treatment development for pediatric trich is to clarify the nature of inhibitory control processes implicated in TTM and to develop a treatment that specifically targets these implicated cognitive processes. Examples of this strategy are found in the increasing availability of translational research that has demonstrated the therapeutic benefits of computerized cognitive training programs (CTPs) in modifying problematic cognitive processes in numerous psychiatric conditions. The objective of this study is to examine the feasibility of CTP for enhancing response inhibition capabilities among individuals with trich, thereby reducing TTM symptoms.

To this end, young individuals aged between 12 and 18 with TTM will be randomly assigned to the CTP condition vs. a wait-list condition. Participants in the CTP condition will receive eight 30-min training sessions over a 4-week period and will be assessed at three time points. Participants in the wait-list will be evaluated at baseline and post-training assessments, and will be allowed to receive the CTP after completing the post-training assessment. Wait-list controls who choose to cross over to the CTP condition will also provide a small replication sample to test the effect of our response inhibition training.

There are three primary implications from this work. First, demonstrating successful enhancement in response inhibition by our proposed CTP is expected to create ample opportunities for clinical research not only on TTM, but also for numerous other psychiatric problems in which poor response inhibition is implicated (e.g., Chronic Skin Picking, Tourette Syndrome, OCD, and ADHD).

This research has the potential to produce a highly cost-efficient self-administered intervention for TTM. Upon establishing efficacy, CTPs may be easily integrated into various contexts, examples include CTPs as an adjunctive intervention to existing behavioral and/or pharmacological treatments, an instrument to identify and help at-risk individuals for preventative training, a stand-alone short-term intervention, and a remote web-based self-help intervention for individuals who have no easy access to treatment resources or are reluctant to seek treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 9 and 17
* A primary diagnosis of Trichotillomania based on DSM-IV criteria (using Trichotillomania Diagnostic Interview)

Exclusion Criteria:

* those who are actively psychotic
* those who have visual impairments that prevent them from performing computer tasks
* those who present developmental disabilities and/or low overall IQ estimated to be below low average (< 79)
* those whose medication status has not been stable
* those who present with past/current substance abuse/dependence problems

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
NIMH Trichotillomania Severity and Impairment Rating Scale | Baseline
  This is one of the most widely clinician-interview based measure designed to assess the severity of hair pulling symptoms during the previous week. We administer this outcome measure at the baseline prior to the intervention.
NIMH Trichotillomania Severity and Impairment Rating Scale | 4 week
  This primary outcome measure will be administered again at 4 week after completing the intervention or after completing the 1-month waiting period.
NIMH Trichotillomania Severity and Impairment Rating Scale | 8 week
  This primary outcome measure will be administered again at 8 week, which is designed for a 1-month follow-up assessment after completing the intervention.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Baseline
  This is a clinician-administered rating scale that is widely used in clinical outcome research to evaluate treatment outcomes with respect to overall levels of severity and improvement.
Clinical Global Impression (CGI) | 4 week
  This measure will be administered at 4 week (after completing the training or 1-month waiting period).
Clinical Global Impression (CGI) | 8 week
  This measure will be administered at 8 week for a 1-month follow-up assessment to examine the longterm effect of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychology Clinic, University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Lee HJ, Espil FM, Bauer CC, Siwiec SG, Woods DW. Computerized response inhibition training for children with trichotillomania. Psychiatry Res. 2018 Apr;262:20-27. doi: 10.1016/j.psychres.2017.12.070. Epub 2018 Jan 5. PMID 29407564